CLINICAL TRIAL: NCT00766467
Title: A Randomized Placebo-Controlled Trial of Armodafinil (Nuvigil) for Fatigue in Patients With Malignant Gliomas Undergoing Radiotherapy With or Without Standard Chemotherapy Treatment
Brief Title: A Randomized Placebo-Controlled Trial of Armodafinil (Nuvigil) for Fatigue in Patients With Malignant Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eudocia Quant Lee, MD (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); University of California, San Diego (Other); Beth Israel Deaconess Medical Center (Other); Cephalon (Industry)
Responsible Party: Sponsor-Investigator, Eudocia Quant Lee, MD, Center for Neuro-Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07-341
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Glioma
Keywords: armodafinil; Nuvigil; fatigue
MeSH Terms: conditions — Glioma; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Armodafinil
  Interventions: Drug: Armodafinil
- Group 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Armodafinil — Taken orally once a day in the morning. Dose will change depending upon level of fatigue
  Other Names: Nuvigil
  Arms: Group 1
Other: Placebo — Placebo taken once a day in the morning
  Arms: Group 2

SUMMARY:
The purpose of this research study is to determine if armodafinil is safe and effective in treating fatigue in patients with malignant gliomas undergoing treatment with radiotherapy plus temodar. Armodafinil is a wakefulness-promoting agent that has been FDA approved for the treatment of excessive daytime sleepiness for a variety of disorders. Armodafinil may also help to reduce radiation-induced fatigue in brain tumor patients.

DETAILED DESCRIPTION:
* Since no one knows for certain if armodafinil improves fatigue in brain tumor patients undergoing radiation therapy, participants will be randomized into one of two study groups. Half of the participants will receive armodafinil and the other half will receive pills with no medicine (placebo). Neither the participant or the study doctor will know what group they are in.
* Participants will be given a study medication-dosing calendar and will take either the study drug or placebo orally once a day for 8 weeks. The dose will be adjusted on days 8,22 or 43, depending upon the level of fatigue. Treatment will begin within 10 days from the radiation start date.
* Participants will be evaluated via documented clinician telephone call and self-administered questionnaires on days 1, 8, 22, 43 and 57.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed malignant glioma including anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma (WHO grade III/IV), glioblastoma multiforme (WHO grade IV) or gliosarcoma. Patients with a grade II astrocytoma, mixed oligo-astrocytoma or oligodendroglioma who are being treated with irradiation are also eligible
* Scheduled to receive irradiation to a total dose of 50-60 Gy. Patients receiving hyperfractionated radiotherapy are also eligible
* KPS of 70% or greater
* Electrolytes within normal institutional limits: BUN and Creatinine < 2.5 x ULN: AST, ALT, Bilirubin < 2.5 x ULN
* Able to swallow medication

Exclusion Criteria:

* History of recent cardiac arrhythmia or unstable angina
* Has taken a psychostimulant or a monoamine oxidase inhibitor on a regular basis within the past 30 days
* Clinically significant untreated sleep apnea
* A history of clinically significant cardiac disease, including a history of recent myocardial infarction, history of unstable angina, history of left ventricular hypertrophy, or a history of ischemic ECG changes, chest pain, arrhythmia, or other clinically significant manifestations of mitral valve prolapse in association with use of CNS stimulants (e.g. caffeine, amphetamines, methylphenidate)
* Uncontrolled hypertension, alcohol or drug abuse, severe headaches, glaucoma, narcolepsy, clinically significant untreated sleep apnea, psychotic disorder or Tourette's syndrome
* Patients taking warfarin for anticoagulation are eligible, but monitoring of prothrombin times is suggested as a precaution
* Hemoglobin level of less then 11 g/dl
* Laboratory evidence of hypothyroidism with an elevated TSH concentration in the blood greater than 5.0 mlU/L
* Current treatment or history of psychotic disorder, bipolar disorder, or anxiety disorder
* Patients with a score of > 28 on the Beck depression inventory consistent with severe depression
* Known hypersensitivity to armodafinil or related compounds
* Patients who have been receiving MAO inhibitors during the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Lee, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - UCSD San Diego, La Jolla, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study activated at Dana-Farber Cancer Institute in August 2008 and was eventually activated at Beth Israel Medical Center , Dartmouth Hitchcock Medical Center, and University of California San Diego. The study closed to new accrual as of April 2014 as the accrual was met.
Pre-assignment Details: Randomization was performed by the Quality Assurance for Clinical Trials office at the Dana Farber Cancer Institute. Patients were randomized in a 1:1 basis to each treatment arm with no stratification.
Groups:
- Armodafinil: Armodafinil: 150mg taken orally once a day in the morning.
- Placebo: Placebo: Taken orally once a day in the morning
Period: Overall Study
Arm/Group | Armodafinil | Placebo
Started | 42 | 39
Initiated Treatment | 39 | 38
Completed | 31 | 31
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 2 | 4
Not completed — Tumor Progression on Study | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Armodafinil: Armodafinil: Taken orally once a day in the morning.
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Placebo | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Continuous [Median (Full Range); unit: years] | 56 [25 to 79] | 54 [19 to 78] | 55 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 24 | 21 | 45
Karnofsky Performance Status (KPS) [Median (Full Range); unit: Units on a scale] — Karnofsky Performance Status ranges from 0 (Dead) to 100 (Normal, no complaints, no evidence of disease) in increments of 10. This was measured at baseline, prior to any treatment on study.
  Units on a scale | 90 [70 to 100] | 90 [70 to 100] | 90 [70 to 100]
Glioma grade [Number; unit: units on a scale] — Glioma is a broad category of brain and spinal cord. Gliomas can be grade I, II, III or IV. For the purposes of this study, Grade II, III, and IV were eligible for enrollment.
  units on a scale
    Grade 2 | 1 | 4 | 5
    Grade 3 | 14 | 12 | 26
    Grade 4 | 25 | 22 | 47
    Grade not defined | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fatigue at Day 43
Description: The primary endpoint was the difference in the 42-day change (baseline vs. day 43) in Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-F scale) between the 2 treatment groups (those patients randomized to receive armodafinil and those randomized to the placebo arm). FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials.5 It consists of the 27-item FACT-G (which assesses QOL based on physical, social/family, emotional, and functional well-being) and the 13-item FACIT-F fatigue subscale (which assesses the impact of fatigue on daily activities). Each item is assessed on a 5-point scale (0 = not at all to 4 = very much). By scoring convention, after appropriate reversal scoring of 11 items, the FACIT-F fatigue subscale (FACIT-fatigue) score ranges from 0 to 52 (lower score indicating more fatigue). A score < 30 indicates severe fatigue.
Time Frame: 43 days
Population: Primary analysis included participants with complete or near complete baseline and day 43 data irrespective of the amount of treatment received.
Measure: Median (80% Confidence Interval); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 31 | 29
units on a scale | -1 [-22 to 48] | -3 [-38 to 22]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.3, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Quality of Life at Days 22, 43 and 56
Description: The effects of treatment on overall health-related quality of life quantified with the general Functional Assessment of Cancer Therapy survey (FACT-G) were measured at baseline, at day 22, at the end of radiation (day 43) and 2 weeks after completion of radiation (day 56). The FACT-G assesses quality of life based on physical, social/family, emotional, and functional well-being. Each item is assessed on a 5-point scale (0 = not at all to 4 = very much). The total FACT-G score can range from 0-108, with higher scores indicating a better quality of life.
Time Frame: baseline, day 22, day 43, and day 56
Population: Analysis included participants with complete or near complete baseline and day 43 data irrespective of the amount of treatment received.
Measure: Median (80% Confidence Interval); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 31 | 29
units on a scale
  FACIT-G (baseline vs day 22) | -1.76 [-45.01 to 24.5] | -4.94 [-45 to 21]
  FACIT-G (baseline vs day 43) | 2.50 [.28 to 25.17] | -2.30 [-58.6 to 20.17]
  FACIT-G (baseline vs day 56) | 1.83 [-40 to 22] | -0.84 [-24 to 16]

3. Secondary Outcome: Number of Grade 3-4 Side Effects at Least Possibly Related to Study Treatment
Description: To assess the side effect profile of armodafinil in patients with malignant gliomas undergoing radiotherapy with or without standard chemotherapy treatment.
Time Frame: 56 days
Population: Grade 3 - 4 events at least possibly related to study treatment.
Measure: Number; unit: number of incidents
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 42 | 39
number of incidents
  Abdominal pain | 1 | 0
  Confusion | 0 | 1
  Dehydration | 1 | 0
  Diarrhea | 1 | 1
  Glaucoma | 0 | 1
  Hyperkalemia | 1 | 0
  Hypokalemia | 1 | 0
  Hypomagnesemia | 1 | 0
  Ileus | 1 | 0
  Insomnia | 1 | 0
  Mood alteration (agitation) | 0 | 1
  Obstruction, cecum | 1 | 0
  Rash | 0 | 1
  Seizure | 1 | 0
  Speech impairment | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from the time armodafinil/placebo was started up to Day 56 contact.
Description: Abnormal laboratory values or diagnostic tests results constitute AEs only if they induce clinical signs or symptoms or require treatment or further diagnostic tests.
Arm/Group | Armodafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 3/42 | 5/39
Other Adverse Events (participants affected / at risk) | 36/42 | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (N=42) | Placebo (N=39)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Obstruction, Cecum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (N=42) | Placebo (N=39)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing-other (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (4) | 3 (3)
Leukocytes (Blood and lymphatic system disorders) | 1 (4) | 5 (11)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 4 (9)
Myelodysplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 2 (3) | 4 (9)
Platelets (Blood and lymphatic system disorders) | 2 (4) | 4 (23)
Hematologic-other (Blood and lymphatic system disorders) | 2 (5) | 5 (13)
Heart block Wolff-Parkinson-White (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac-other (Cardiac disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 17 (20) | 15 (20)
Fever w/o neutropenia (General disorders) | 2 (3) | 1 (1)
Insomnia (General disorders) | 13 (17) | 11 (15)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Constitutional, other (General disorders) | 3 (4) | 0 (0)
Coagulation-other (Investigations) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin-other (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (2)
Cushingnoid appearance (Endocrine disorders) | 1 (1) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 7 (7)
Constipation (Gastrointestinal disorders) | 10 (10) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Teeth development (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (4) | 1 (1)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (17) | 11 (11)
Taste disturbance (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (4)
GI-other (Gastrointestinal disorders) | 1 (1) | 1 (2)
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection w/ gr3-4 neut, oral cavity (Infections and infestations) | 1 (1) | 0 (0)
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 0 (0) | 1 (1)
Infection Gr0-2 neut, paranasal (Infections and infestations) | 1 (1) | 0 (0)
nfection Gr0-2 neut, urinary tract (Infections and infestations) | 0 (0) | 1 (2)
nfection Gr0-2 neut, wound (Infections and infestations) | 1 (1) | 0 (0)
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 (0) | 1 (1)
Infection-other (Infections and infestations) | 0 (0) | 1 (1)
Edema head and neck (General disorders) | 1 (1) | 0 (0)
Edema limb (General disorders) | 1 (1) | 1 (1)
Lymphatics-other (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
ALT, SGPT (Investigations) | 1 (1) | 4 (4)
AST, SGOT (Investigations) | 0 (0) | 1 (1)
Hypercalcemia (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Investigations) | 3 (3) | 2 (6)
Hypoglycemia (Investigations) | 1 (1) | 0 (0)
Lipase (Investigations) | 1 (1) | 0 (0)
Hypomagnesemia (Investigations) | 1 (1) | 0 (0)
Hyperkalemia (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Investigations) | 1 (3) | 0 (0)
Hyponatremia (Investigations) | 1 (1) | 0 (0)
Metabolic/Laboratory-other (Investigations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (5) | 0 (0)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nonneuropathic lower extr muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nonneuropathic upper extr muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nonneuropathic left-side muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
CNS necrosis/cystic progression (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 7 (9) | 6 (7)
Memory impairment (Nervous system disorders) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 12 (13) | 4 (5)
Depression (Psychiatric disorders) | 2 (2) | 4 (4)
Neuropathy CN II vision (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy-motor (Nervous system disorders) | 1 (1) | 3 (5)
Neuropathy-sensory (Nervous system disorders) | 1 (1) | 3 (3)
Seizure (Nervous system disorders) | 2 (3) | 1 (3)
Speech impairment (Nervous system disorders) | 2 (5) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Neurologic-other (Nervous system disorders) | 3 (4) | 7 (7)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Vision-blurred (Eye disorders) | 2 (2) | 2 (2)
Ocular-other (Eye disorders) | 1 (1) | 0 (0)
Abdomen, pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Back, pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental/teeth/peridontal, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 15 (23) | 11 (13)
Joint, pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (3)
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5)
Neck, pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Pain- other (General disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal - other (Renal and urinary disorders) | 2 (2) | 0 (0)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less